CLINICAL TRIAL: NCT05361135
Title: 18-fluorodeoxyglucose Positron Emission Tomography/Computed Tomography in Staphylococcus Aureus Bacteraemia (Bacteremia/Bloodstream Infection); an International, Multicentre, Randomised Control Trial
Brief Title: 18-fluorodeoxyglucose Positron Emission Tomography/Computed Tomography in S. Aureus Bacteraemia
Acronym: PET-SAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: King's College London (Other); University of Melbourne (Other); Menzies School of Health Research (Other); Olivia Newton-John Cancer Research Institute (Other); Alliance Medical, UK (Unknown); Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PET-SAB
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Staphylococcus Aureus Bacteremia; Staphylococcus Aureus Septicemia; Sepsis Bacterial; Bloodstream Infection; Staph Sepsis; Staphylococcus Aureus Infection; Sepsis
Keywords: Staphylococcus; Staphylococcus Aureus Bacteremia; Staphylococcus Aureus Septicemia; Sepsis; Sepsis Bacterial; Staph Sepsis; Staphylococcus Aureus Infection; Bloodstream Infection; Staphylococcus Aureus Bacteraemia; PET; PET/CT; PET-CT; Positron Emission Tomography; Positron Emission Tomography/Computed Tomography; Diagnostic Imaging
MeSH Terms: conditions — Sepsis; Staphylococcal Infections | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PET/CT (Experimental): Enhanced imaging with PET/CT
  Interventions: Diagnostic Test: PET/CT
- Routine Imaging (No Intervention): Standard of Care Imaging

INTERVENTIONS:
Diagnostic Test: PET/CT — Enhanced imaging with PET/CT
  Other Names: PET-CT
  Arms: PET/CT

SUMMARY:
Having bacteria in the blood can be very dangerous. This is called bacteraemia (or bacteremia) or bloodstream infection. It can lead to problems across the whole body, which is what happens in sepsis. Bacteria called Staphylococcus aureus (S. aureus) cause one kind of bacteraemia. Up to a third of people with this condition die within three months, even with antibiotics. One reason for such severe problems is that the bacteria can spread almost anywhere in the body, and hide in places where they are very hard to find. When people with S. aureus bacteraemia come into hospital and have had antibiotics, doctors sometimes cannot tell if they still have an infection source (called a 'focus') hiding in their body. The focus can be like an abscess and may need removing or the pus draining out. A focus might be obvious, if there is pain or swelling, or it might be hidden and deep. If these 'foci' can be found, then doctors can treat them and this helps to cure patients.

To improve survival for patients with these life-threatening infections, it is vital that doctors find the focus of S. aureus bacteraemia as quickly as possible. However, the research team do not know the best way to do this. Most patients with S. aureus bacteraemia have a chest X-ray and a scan of the heart valves. Patients may go to the scanning department lots of times while doctors try to work out where these foci are. This is uncomfortable and takes a lot of time. In about 1 in 5 cases the doctors still cannot find the focus. This is very worrying for patients, their relatives and doctors.

This study has been designed by researchers, doctors and patient advocates. It aims to work out if fewer patients may die when a specific type of scan called a 'PET/CT' is done quickly, because it finds more foci. To do this the team plan to do a clinical trial in patients with S. aureus bacteraemia. Half of the patients will receive the usual tests that patients currently get and the other half will receive an extra scan as soon as possible. The patients will be chosen randomly (like the flip of a coin) to go into one of the 2 groups. A year into the trial, an independent committee will check the results to make sure the extra scan is finding more foci. If this is the case, the trial will carry on. At the end of the study, we will share the results globally. The findings are expected to change the way this dangerous condition is managed, so patients do better.

DETAILED DESCRIPTION:
Staphylococcus aureus (S. aureus) bacteraemia/bloodstream infection (SAB) is associated with deep foci in a high proportion of cases, through local or haematogenous spread or seeding. Detecting infectious foci in SAB is a prerequisite to source control, which is critical to improving outcomes. However, in up to 1 in 5 cases no focus can be found, and in others additional foci may be missed. When the foci are not found, this is associated with higher mortality.

Positron emission tomography/computed tomography (usually with 18-fluorodeoxyglucose (FDG), denoted PET/CT) is increasingly available worldwide. The role of PET/CT to rapidly detect deep infectious foci in SAB is becoming clearer with increasing use. The European Medicines Agency licensed FDG for use in PET/CT investigation of bacteraemia based on observational studies. Single-centre observational studies have found PET/CT detected infectious foci in the majority of cases of SAB. A prospective matched cohort study found a suggestion of improved survival with the use of PET/CT, though the rates of solid malignancies and nosocomial infection were higher in the control group. This is a multi-centre randomised controlled trial (RCT) of PET/CT in SAB.

The hypothesis is that PET/CT within 14 days of platform entry to SNAP enables the detection of new foci of infection leading to improved clinical outcomes.

The null hypothesis is that a composite of 90-day all-cause mortality or microbiological relapse or microbiological treatment failure will not be changed by early PET/CT in SAB.

Primary outcome:

A composite of 90-day all-cause mortality or microbiological relapse or microbiological treatment failure 90 days after platform entry.

Secondary outcomes:

The detection of new foci between 0 and 90 days after platform entry. The presence of new foci will be determined by the site investigator and can incorporate clinical, radiological, microbiological and pathological findings.

The presence of new foci will be determined by the site investigator and can incorporate clinical, radiological, microbiological and pathological findings.

All cause mortality at 90 days after platform entry Duration of survival censored at 90 days after platform entry. Length of stay of acute index inpatient hospitalisation for those surviving until hospital discharge (excluding or including HITH/COPAT/OPAT/rehab) truncated at 90 days after platform entry Time to being discharged alive from the total index hospitalisation (excluding or including HITH/COPAT/OPAT/rehab) truncated at 90 days after platform entry.

Microbiological treatment failure defined as positive sterile site culture for S. aureus between 14 and 90 days after platform entry.

Total radiation exposure Patient Eligibility Criteria Inclusion criteria: Adult (≥18 years of age) and consented to the SNAP platform. Agrees to PET/CT.

Exclusion criteria:

Contraindication to PET/CT (including pregnancy/breast-feeding) PET/CT in the last 7 days or already planned to occur in the next 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age)
* Staphylococcus aureus complex grown from ≥1 blood culture
* Symptoms of S. aureus bloodstream infection
* Admitted to a participating hospital at the time of eligibility assessment . Agrees to PET/CT

Exclusion Criteria:

* Contraindication to PET/CT (including pregnancy/breast-feeding)
* PET/CT in the last 7 days or already planned to occur in the next 7 days
* Treating team deems enrolment in the study is not in the best interest of the patient
* Treating team believes that death is imminent and inevitable
* Patient is for end-of-life care and PET/CT is considered not appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days
  All cause mortality- Number of participants who are no longer alive at day 90

SECONDARY OUTCOMES:
Total antibiotic days | 90 days
  Total number of days of antibiotic and type (IV or oral delivery) per participant measured at day 90
Source control | Time to hospital total discharge [up to 90 days from platform entry]
  Control of infection sites through surgery, drainage and other procedures- Number of participants who receive these procedures and number of participants in whom these procedures are not completed but infectious foci remain
Number of participants with a change in the planned management strategy | Time to hospital total discharge [up to 90 days from platform entry]
  Number of participants with a change in the planned management strategy by date of total hospital discharge (including OPAT)
Length of Stay | 90 days
  Length of stay of acute index inpatient hospitalisation for participants surviving until hospital discharge
Microbiological failure and relapse | From 14 to 90 days
  Microbiological treatment failure and relapse defined as positive sterile site culture for S. aureus from a participant
Adverse events including total radiation exposure | 90 days
  Total radiation exposure to the participant and serious adverse events
Diagnosis of new infectious foci | Up to 90 days after platform entry
  Detection of Deep Foci of Infection in the participant (location). The presence of deep foci will be determined by the site investigator and can incorporate clinical, radiological, microbiological and pathological findings.
Composite of 90-day all-cause mortality or microbiological relapse or microbiological treatment failure. | Up to 90 days after platform entry
  Number of participants with a composite of 90-day all-cause mortality or microbiological relapse or microbiological treatment failure. Microbiological relapse is defined as a positive blood culture for S. aureus at least 72 hours after a preceding negative culture. Microbiological treatment failure is defined as a positive sterile-site culture for S. aureus of the same antibiotic resistance as the index isolate at least 21 days after platform entry.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Goodman, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: Yes
This will be determined with the protocol. It is will be open but would need to protect patient identifiable data.
Supporting Information: Study Protocol, SAP
Time Frame: To be determined
Access Criteria: Open access Study Protocol